CLINICAL TRIAL: NCT01086761
Title: A Phase I/II, Open-label, Non-controlled, Escalating Dose, Multicentre Clinical Trial Evaluating the Safety, Preliminary Efficacy, and Pharmacokinetics of MP0112 Injected Intravitreally in Patients With Wet Age Related Macular Degeneration (AMD)
Brief Title: Study of MP0112 Intravitreal Injection in Patients With Wet Age Related Macular Degeneration
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a company decision following completion of Part A.
Sponsor: Allergan (Industry)
Collaborators: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP0112-CP01
Record Dates: First submitted 2010-03-09; First posted 2010-03-15 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Wet Age-Related Macular Degeneration
MeSH Terms: interventions — MP0112

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- MP0112 (0.04 mg) (Experimental): Single 0.04 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112
- MP0112 (0.15 mg) (Experimental): Single 0.15 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112
- MP0112 (0.4 mg) (Experimental): Single 0.4 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112
- MP0112 (1.0 mg) (Experimental): Single 1.0 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112
- MP0112 (2.0 mg) (Experimental): Single 2.0 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112
- MP0112 (3.6 mg) (Experimental): Single 3.6 mg intravitreal injection of MP0112 in the study eye.
  Interventions: Biological: MP0112

INTERVENTIONS:
Biological: MP0112 — Single intravitreal injection of MP0112 in the study eye.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of MP0112 (a novel, potentially long acting VEGF inhibitor) in patients with wet Age Related Macular Degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and angiographic evidence of active primary progressive subfoveal choroidal neovascularisation (CNV), including juxtafoveal lesions that affect the fovea on FA in the study eye that is at least 50% of the total lesion area
* ETDRS best-corrected visual acuity of: 20/40 to 20/320 in the study eye at 4 meters
* Male or female age > 50 years
* Written informed consent prior to any study procedures
* Willing, committed, and able to return for ALL clinic visits and complete all study-related procedures.

Exclusion Criteria:

* Prior treatment with anti-VEGF therapy in the study eye, including bevacizumab, ranibizumab, or pegaptanib, as well as photodynamic therapy with verteporfin
* Any prior or concomitant therapy with another investigational agent to treat neovascular AMD in the study eye, except dietary supplements or vitamins
* Subfoveal thermal laser therapy, external-beam radiation therapy, or transpupillary thermotherapy in the study eye
* Extrafoveal laser coagulation treatment within 12 weeks prior to Baseline in the study eye
* Total lesion size > 20mm2 (including blood, scars and neovascularization) as assessed by FA in the study eye
* Subretinal hemorrhage that is either 50% or more of the total lesion area, or if the blood is under the fovea and is 2.54mm2 or more in size in the study eye
* Scar or fibrosis, making up > 50% of total lesion in the study eye
* Scar, fibrosis, or atrophy involving the center of the fovea
* Presence of retinal pigment epithelial tears or rips
* History of any vitreous hemorrhage within 4 weeks prior to Visit 1 or current hemorrhage in the study eye
* Presence of other causes of CNV, including pathologic myopia (spherical equivalent of -8 diopters or more negative, or axial length of 25 mm or more), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, or multifocal choroiditis in the study eye
* History or clinical evidence of diabetic retinopathy, diabetic macular oedema or any other vascular disease affecting the retina, other than AMD, in either eye
* Prior vitrectomy in the study eye
* History of retinal detachment or treatment or surgery for retinal detachment in the study eye
* Ocular surgery (including cataract removal) in the study eye within 3 months of enrolment
* Active intraocular inflammation (grade trace or above) in the study eye
* History of allergy to any components of the study drug or diagnostic devices, such as fluorescein
* Advanced glaucoma or intraocular pressure above 22 mmHg in the study eye despite treatment
* Inability to obtain fundus photographs or fluorescein angiogram of sufficient quality to be analyzed and graded by the central reading center
* History of idiopathic or autoimmune-associated uveitis in either eye
* Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or absence of the posterior capsule in the study eye
* Presence of a non-healing wound, ulcer, fracture or any other medical condition associated with bleeding
* Use of antimitotic or antimetabolite therapy within 30 days or 5 elimination half-lives of enrolment
* Premenopausal women
* Any disorder or condition that contraindicates the use of an investigational drug
* Participation in another investigational drug study within 3 months of enrolment
* Uncontrolled hypertension
* Previous stroke within 12 months of study entry
* Systemic treatment with any anti-VEGF drug
* Current treatment for active systemic infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Czechia (3):
  - Fakultni Nemocnice Brno, Brno, Czech
  - Fakultni Nemocnice Olomouc, Olomouc, Czech
  - Ustrendi Vojenska Nemocnice, Prague, Czech
- France (4):
  - Hopital Intercommunual de Creteil, Créteil, Creteil
  - Centre Rabelais, Lyon, Lyon
  - Centre Paradis-Monticelli, Marseille, Marseille
  - Hopitaux Universitaires, Strasbourg, Strasbourg
- Inselspital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Souied EH, Devin F, Mauget-Faysse M, Kolar P, Wolf-Schnurrbusch U, Framme C, Gaucher D, Querques G, Stumpp MT, Wolf S; MP0112 Study Group. Treatment of exudative age-related macular degeneration with a designed ankyrin repeat protein that binds vascular endothelial growth factor: a phase I/II study. Am J Ophthalmol. 2014 Oct;158(4):724-732.e2. doi: 10.1016/j.ajo.2014.05.037. Epub 2014 Jun 5. PMID 24907435

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | MP0112 (1.0 mg) | MP0112 (2.0 mg) | MP0112 (3.6 mg)
Started | 9 | 7 | 6 | 6 | 4 | 0
Completed | 9 | 7 | 6 | 6 | 4 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | MP0112 (1.0 mg) | MP0112 (2.0 mg) | Total
Number analyzed (Participants) | 9 | 7 | 6 | 6 | 4 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.2 (6.3) | 78.6 (3.2) | 77.5 (6.0) | 79.0 (3.0) | 77.8 (9.4) | 78.3 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 3 | 3 | 2 | 21
  Male | 1 | 2 | 3 | 3 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximal Tolerated Dose (MTD) Following a Single Injection
Description: MTD was defined as one dose level below the lower of the dose level in which a severe (sight-threatening) drug-related Adverse Event occurred or the dose level at which more than 2 patients experienced a moderate ocular (eye) drug-related toxicity.
Time Frame: 16 weeks
Population: All treated participants.
Measure: Number; unit: mg
Groups:
- MP0112: Single intravitreal injection of MP0112 in the study eye of one of the following doses: 0.04 mg, 0.15 mg, 0.4 mg, 1.0 mg or 2.0 mg.
Arm/Group | MP0112
Number analyzed (Participants) | 32
mg | 1.0

2. Secondary Outcome: Percentage of Participants With Stable or Improved Best Corrected Visual Acuity (BCVA)
Description: BCVA was measured using an eye chart and was reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye at Baseline and Week 4. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the letters read correctly on the eye chart the better the vision. Stable or Improved BCVA was defined as a loss of <15 letters read correctly compared to Baseline.
Time Frame: Baseline, Week 4
Population: All treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | MP0112 (1.0 mg) | MP0112 (2.0 mg)
Number analyzed (Participants) | 9 | 7 | 6 | 6 | 4
Percentage of participants | 100 | 100 | 100 | 83 | 75

3. Secondary Outcome: Change From Baseline in Central Area Retinal Thickness
Description: Optical Coherence Tomography (OCT), a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina, was performed in the study eye after pupil dilation at Baseline and Week 4. A negative change from Baseline indicated improvement (less retinal thickness). A positive change from Baseline indicated worsening (definite retinal thickening).
Time Frame: Baseline, Week 4
Population: All treated participants.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | MP0112 (1.0 mg) | MP0112 (2.0 mg)
Number analyzed (Participants) | 9 | 7 | 6 | 6 | 4
μm
  Baseline | 353.0 (79.3) | 338.0 (69.7) | 367.2 (213.5) | 333.3 (79.4) | 375.3 (69.3)
  Change from Baseline at Week 4 | 21.6 (118.2) | 10.1 (102.8) | -39.8 (72.4) | -95.0 (91.2) | -99.0 (35.5)

4. Secondary Outcome: Area of Leakage as Measured by Fluorescein Angiography
Description: Fluorescein angiography (FA) is a technique for examining the circulation of the retina (and detecting any leakage) using a dye-tracing method. Photographs are taken with a specialized low-power microscope with an attached camera designed to photograph the interior of the eye, including the retina and optic disc. FA was performed on the dilated study eye 10 minutes after fluorescein application at Baseline and Week 4. A lower number indicated a smaller area of leakage.
Time Frame: Baseline, Week 4
Population: All treated participants.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | MP0112 (1.0 mg) | MP0112 (2.0 mg)
Number analyzed (Participants) | 9 | 7 | 6 | 6 | 4
mm^2
  Baseline | 15.0 (4.0) | 9.5 (3.0) | 12.8 (5.9) | 8.4 (4.0) | 10.2 (7.5)
  Week 4 (n=9,7,6,6,3) | 4.1 (4.9) | 2.6 (3.5) | 2.4 (3.8) | 1.0 (2.4) | 0.0 (0.0)

5. Secondary Outcome: Area of Lesion as Measured by Fluorescein Angiography
Description: Fluorescein angiography (FA) is a technique for examining the circulation of the retina (and detecting any leakage) using a dye-tracing method. Photographs are taken with a specialized low-power microscope with an attached camera designed to photograph the interior of the eye, including the retina and optic disc. FA was performed on the dilated study eye after fluorescein application at Baseline and Week 4. A lower number indicated a smaller lesion area.
Time Frame: Baseline, Week 4
Population: All treated participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | MP0112 (1.0 mg) | MP0112 (2.0 mg)
Number analyzed (Participants) | 9 | 7 | 6 | 6 | 4
mm^2
  Baseline | 13.9 (3.9) | 8.0 (3.6) | 12.1 (6.9) | 9.5 (4.4) | 10.9 (7.9)
  Week 4 (n=9,6,6,6,2) | 8.3 (4.8) | 6.2 (3.9) | 6.8 (4.1) | 7.3 (4.6) | 11.7 (6.1)

6. Secondary Outcome: Maximum Serum Concentration (Cmax) of MP0112 at Day 3
Description: Blood samples were collected for MP0112 levels on Day 3. The serum samples (liquid portion of the blood after cells and clotting factors were removed) were sent to a laboratory and were analyzed for MP0112 levels using an enzyme-linked immunosorbent assay. Maximum concentration at Day 3 was calculated.
Time Frame: Day 3
Population: Pharmacokinetic (PK) Population included all treated participants with PK data.
Measure: Number; unit: Nanomolar (nM)
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | MP0112 (1.0 mg) | MP0112 (2.0 mg)
Number analyzed (Participants) | 9 | 7 | 6 | 6 | 4
Nanomolar (nM) | NA (NA) — Result is below the lower limit of quantitation of the laboratory test: <0.3 nM. | NA (NA) — Result is below the lower limit of quantitation of the laboratory test: <0.3 nM. | NA (NA) — Result is below the lower limit of quantitation of the laboratory test: <0.3 nM. | 0.5 | 1.0

7. Secondary Outcome: Number of Participants With Positive Binding Anti-MP0112 Antibodies
Description: Blood samples were collected Pre-treatment (Baseline) and Weeks 4, 8 and 12. Samples were analyzed for Anti-MP0112 antibodies using an enzyme-linked immunosorbent assay.
Time Frame: 12 weeks
Population: Safety Population included all treated participants.
Measure: Number; unit: Participants
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | MP0112 (1.0 mg) | MP0112 (2.0 mg)
Number analyzed (Participants) | 9 | 7 | 6 | 6 | 4
Participants | 0 | 1 | 3 | 1 | 3

ADVERSE EVENTS:
Arm/Group | MP0112 (0.04 mg) | MP0112 (0.15 mg) | MP0112 (0.4 mg) | MP0112 (1.0 mg) | MP0112 (2.0 mg)
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 0/6 | 0/6 | 1/4
Other Adverse Events (participants affected / at risk) | 8/9 | 7/7 | 6/6 | 4/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP0112 (0.04 mg) (N=9) | MP0112 (0.15 mg) (N=7) | MP0112 (0.4 mg) (N=6) | MP0112 (1.0 mg) (N=6) | MP0112 (2.0 mg) (N=4)
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP0112 (0.04 mg) (N=9) | MP0112 (0.15 mg) (N=7) | MP0112 (0.4 mg) (N=6) | MP0112 (1.0 mg) (N=6) | MP0112 (2.0 mg) (N=4)
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 7 | 7 | 5 | 2 | 2
Anterior chamber inflammation (Eye disorders) | 0 | 1 | 1 | 2 | 1
Anterior chamber cell (Eye disorders) | 0 | 0 | 1 | 0 | 2
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0
Corneal epithelium defect (Eye disorders) | 0 | 0 | 0 | 0 | 1
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Macular cyst (Eye disorders) | 1 | 0 | 0 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ocular toxicity (Eye disorders) | 0 | 0 | 0 | 0 | 1
Pseudoendophthalmitis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal neovascularisation (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0
Subretinal fibrosis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vitreal cells (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vitreous opacities (Eye disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0
Intraocular pressure decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Vitritis (Eye disorders) | 0 | 1 | 0 | 2 | 1
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.